CLINICAL TRIAL: NCT05660993
Title: Multicenter Study of Safety and Efficacy of PET-adapted Treatment With Nivolumab, Bendamustine, Gemcitabine, Vinorelbine (Nivo-BeGEV) in Patients With Relapsed/Refractory Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, Vice-director Nathional Medical Research Center for Hematology Moscow Russia, National Research Center for Hematology, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: r/r cHL-2022
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Hodgkin Lymphoma
Keywords: PET-adapted Treatment; Relapsed/Refractory Hodgkin Lymphoma; Nivolumab; BeGEV
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Experimental): Patients will receive for a maximum of 4 cycles of nivolumab 3 mg/kg on day 0 BeGEV , with subsequent assessment of response by PET-CT. Patients with CR after 2 cycles Nivo-BeGEV will proceed to ASCT.
  Patients with <CR after 2 cycles of a combination Nivo-BeGEV, with subsequent PET-CT assessment, will receive an additional 2 cycles Nivo-BeGEV. Patients with CR after 4 cycles Nivo-BeGEV will proceed to ASCT.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Drug: Nivolumab Schedule: Nivolumab 3 mg/kg on day 0 of the Nivo-BeGEV or a maximum of 4 cycles Drug: Bendamustine
  Schedule:
  Day 2: Bendamustine 90mg/mq Day 3: Bendamustine 90mg/mq for a maximum of 4 cycles Other Name: Ribomustin
  Drug: Gemcitabine Day 1: Gemcitabine 800mg/mq, Day 4: Gemcitabine 800mg/mq for a maximum of 4 cycles Other Name: Gemzar
  Drug: Vinorelbine Day 1 Vinorelbine 20mg/mq for a maximum of 4 cycles Other Name: Navelbine

SUMMARY:
Nivolumab is an anti-PD-1 antibody highly effective in patients with relapsed/refractory classical Hodgkin lymphoma. A PET-adapted regimen of nivolumab combined with salvage therapy was shown to induce high response rates and favorable progression-free survival as a bridge to autologous stem cell transplantation, allowing to omit salvage chemotherapy in a substantial proportion of r\r cHL patients. This study evaluates the safety and efficacy of PET-adapted treatment of nivolumab at the 3 mg/kg in combination with Bendamustine, Gemcitabine, Vinorelbine (Nivo-BeGEV) in patients with relapsed/refractory Hodgkin Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed Hodgkins lymphoma
* Relapsed or refractory disease after the first line of treatment
* Age 18-70 years old
* Ejection fraction greater than 50%
* ECOG 0-2 status
* Signed informed consent
* No severe concurrent illness

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Severe organ failure: creatinine more than 2 norms; ALT, AST more than 5 norms; bilirubin more than 1.5 norms
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign an informed consent
* Active or prior documented autoimmune disease requiring systemic treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
1. Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 Toxicity parameters based on NCI CTCAE 4.03 grades | 12 months
2. Overall Response Rate (ORR) Overall response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by LYRIC and Lugano 2014 criteria | 12 months

SECONDARY OUTCOMES:
1. Duration of Response (DOR) | 24 months
Overall Survival (OS) | 24 months
Progression-Free Survival (PFS) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Parovichnikova,, MD,PhD, Study Director — Nathional Medical Research Center for Hematology Moscow Russia 125167
Locations (1):
- National Research Center for Hematology, Moscow, Russia